CLINICAL TRIAL: NCT02544685
Title: Prevention of Febrile Neutropenia in Pediatric Cancer Patients by Lactobacillus Rhamnosus GG and Bifidobacterium Animalis Subspecies. Lactis BB-12 in Combination With Inulin and Oligofructose
Brief Title: Prevention of Febrile Neutropenia by Synbiotics in Pediatric Cancer Patients
Acronym: FENSY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: S&D Pharma SK s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2015-08-16; First posted 2015-09-09 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Febrile Neutropenia; Neutropenia; Infection in an Immunocompromised Host; Cancer
Keywords: Febrile neutropenia; Synbiotic; Probiotic; Prebiotic; Safety; Cancer; Oncology; Chemotherapy; Symbiotic
MeSH Terms: conditions — Febrile Neutropenia; Neutropenia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synbiotics group (Active Comparator): Interventions: administration of Probio-Fix Inum + Beneo Synergy 1
  Start of prophylaxis: 5 days before or 2 days after starting chemotherapy
  Prophylaxis duration: 3 months
  Interventions: Dietary Supplement: Probio-Fix Inum; Dietary Supplement: Beneo Synergy 1
- Placebo group (Placebo Comparator): Interventions: administration of placebo
  Start: 5 days before or 2 days after starting chemotherapy
  Duration: 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probio-Fix Inum — Dose of Probio-Fix Inum: 1 capsule daily first 14 days + 1 capsule twice daily for the rest of prophylaxis duration
  Probio-Fix Inum: each capsule contains 2.7 billion lyophilized probiotic bacteria Lactobacillus rhamnosus GG, LGG, American Type Culture Collection (ATCC) 53103 and Bifidobacterium animalis subspecies. lactis BB-12 Chr. Hansen Beneo Synergy 1: oligofructose-enriched inulin
  Arms: Synbiotics group
Dietary Supplement: Beneo Synergy 1 — Dose of Beneo Synergy 1: depends on the age of the patient (full dose variation: 0,2g/100ml milk formula - 12g/daily), gradually increased as tolerated by the patient every 2-3 days in first 8-12 days
  Arms: Synbiotics group
Other: Placebo — Same dosage regimen as active drugs
  Arms: Placebo group

SUMMARY:
Febrile neutropenia (FN) is a major life-threatening treatment complication in cancer patients undergoing intensive chemotherapy. Endogenous flora is considered to be one of the main sources of infections during neutropenia. Competitive inhibition of gut mucosal colonization by pathogenic microorganisms using synbiotics could represent one of the potential options for its prevention. Synbiotics represent combination of two components: probiotics and prebiotics. Probiotics are live microorganisms, which in form of drugs or food supplements administered at a sufficient dose help to maintain health beneficial microbial balance in the digestive tract of a human or other host. Prebiotics are food ingredients nondigestible for our digestive enzymes, but can be fermented by bacteria in our bowel and this way selectively stimulate growth or activity of specific saccharolytic bacterial strains. These changes in composition of our microflora may bring benefits on host well-being and health. Based on the results of human and animal studies, probiotics probably can not only decrease the level of gut colonisation with pathogenic bacteria, but may also lead to reduction in the duration of neutropenia, accelerate the restitution of the intestinal mucosa and boost immunity. Despite a significant number of studies on probiotics still only little evidence of their safety especially in immunocompromised patients is available.

To help find new options for increasing quality of healthcare for children cancer patients and also to evaluate safety of this new approach investigators designed double-blinded placebo controled multicenter study aimed to decrease the number of febrile episodes using prevention with synbiotic.

DETAILED DESCRIPTION:
Febrile neutropenia (FN) is a major complication in cancer patients undergoing intensive chemotherapy. Endogenous flora is considered to be one of the main sources of infections in neutropenic patients. The first step in infection process is colonization of the intestine by pathogenic bacteria with their subsequent translocation through the intestinal mucosa and systemic dissemination.

The alterations of the intestinal flora occurs due to chemotherapy and also due to the use of broad spectrum antibiotics, which suppresses anaerobic growth of the normal gut flora leading to a damage of colonization resistance. Competitive inhibition of gut mucosal colonization by pathogenic micro-organisms using synbiotics could represent one of the potential options for the prevention of febrile neutropenia in cancer patients. Compared with the existing selective bowel decontamination with quinolones and/or trimethoprim-sulfamethoxazole, investigators may expect also reduction of the incidence of fungal and Gram-positive infections due to changes in the intestinal microflora. Based on the results of animal studies, probiotics could probably also lead to a reduction in the duration of neutropenia and boost immunity.

Synbiotics represent combination of two components: probiotics and prebiotics. Probiotics are live microorganisms, which in form of drugs or food supplements administered at a sufficient dose help to maintain health beneficial microbial balance in the digestive tract of a human or other host. Prebiotics are food ingredients nondigestible for our digestive enzymes, but can be fermented by bacteria in our bowel and this way selectively stimulate growth or activity of specific saccharolytic bacterial strains.

Lactic acid bacteria are currently widely used in prevention and treatment of certain infectious diseases. They stimulate the immune system, compete for substrate with pathogenic bacteria, produce bacteriocins, competitively inhibit bacterial adhesion sites, increase the transepithelial resistance and bind some mutagens.

Current evidence supporting probiotic use as adjunctive therapy to anticancer treatment is limited, especially in cancer patients treated with chemotherapy. Some of the reports support their beneficial effects on certain aspects of toxicity related to chemotherapy and radiation therapy; however, large properly designed clinical trials are needed to assess their real position as a part of anticancer treatment.

Eleven studies in cancer patients were included in meta-analysis to assess efficacy of probiotics. Results show that probiotics may reduce the severity and frequency of diarrhoea in patients with cancer and may reduce the requirement for anti-diarrhoeal medication, but still more studies are needed to assess the true effect. The importance of probiotics in the treatment of acute diarrhea is supported by meta-analysis of 34 randomized placebo-controlled studies, which showed significant reduction in diarrhea incidence with better effect especially in the pediatric group. Most of these studies were performed with the probiotic strain Lactobacillus rhamnosus GG (LGG). The duration of rotavirus diarrhea in children and diarrhea in immunocompromised HIV-positive patients was significantly shortened after administration of certain strains of Lactobacilli resp. Saccharomyces boulardii.

Investigators can find only anecdotal reports about use of probiotics in patients with neutropenia. In experimental models with cyclophosphamide-treated mice preventive treatment with immunomodulatory lactobacilli was successfully used to protect against myelosuppression and immunosuppression. Lactobacilli were able to induce an early recovery of neutrophils in blood, improve phagocytic cells recruitment to infectious sites and increase the resistance against the opportunistic pathogen C. albicans. In another similar study administration of heat-inactivated strain of Enterococcus faecalis shortened the duration of cyclophosphamide-induced neutropenia and speeded up the restitution of neutrophil count. The important feature of the lactic acid bacteria is ability to produce fatty acids with short chain, which is an important metabolite for colonocytes and this way they may participate in the faster restitution of the mucosa after chemotherapy.

Probiotics fall into the category of organisms classified as "generally regarded as safe". The safety concerns with probiotic administration in cancer patients are related mainly to risk of infection caused by probiotic bacteria and transfer of antibiotics resistance.

Many probiotics strains are naturally resistant to antibiotics, but majority of this resistance is intrinsic (chromosomally encoded) and therefore nontransmissible. This could be a danger, when probiotics become infectious agents, on the other hand probiotic strains with intrinsically antibiotic-resistance may benefit patients, whose normal intestinal microflora has become greatly reduced or unbalanced due to the administration of various antimicrobial agents. For some strains (e.g. LGG) the plasmid-free status was proven, but at the same time it was shown, that some strains may carry potentially transmissible plasmid-encoded antibiotic resistance genes, which could lead to the formation of new antibiotic-resistant pathogens. Therefore, one of the key requirement for probiotic strains is that they should not carry transmissible antibiotic resistance genes.

Despite the fact, that the incidence of infections caused by lactic acid bacteria is extremely low, there exists certain risk, that they can become pathogenic. In case reports probiotics are mentioned as causing local infections such as chest infections, digestive tract infections, urinary tract infections, and meningitis. Though reported lactobacilli bacteremia are very unusual and rare in the pediatric population. They were naturally more often observed in immunocompromised patients, such as in patients with bone marrow transplantation or in patients with AIDS, which also demonstrates low-virulency of these strains. Moreover, clinical isolates of L. rhamnosus captured in these cases had some significant phenotypical differences in one or more properties associated with virulence compared to those, which are used as probiotic strains. Concerns of iatrogenic infection are one of the main reasons for limited experience with administration of probiotics in granulocytopenic patients. In addition, due to chemotherapy it comes not only to neutropenia but also to local affection of gut mucosa and therefore hypothetically arise the possibility of bacterial translocation. This phenomenon is caused by a defective intestinal barrier, immunosuppression and also gut prematurity. It was described as the passage of viable indigenous bacteria from the gastrointestinal tract to extraintestinal sites and may result in the transfer of bacteria to other organs, thereby potentially causing bacteremia, septicemia, and multiple organ failure. However, evidence from animal model studies suggests that there is actually a reduction in the translocation of other bacteria when probiotics are given, as opposed to the transmigration of probiotic bacteria into the bloodstream.

The concerns around bacteraemia/fungaemia or blood culture growth are significant in cancer patients, but this risk needs to be considered alongside any potential benefit. Systematic review including 17 studies with cancer patients identified only five such case reports of the 756 cases described consuming probiotics. Moreover such cases were noted also in patients not known to be consuming probiotics. In addition, there is no evidence from population based studies of any increased risk of bacteremia or endocarditis due to probiotics and their incidence still remained extremely low despite current widespread use of probiotic. Even findings of some small studies in groups of specific immunocompromised patients (e.g., patients with HIV infection) support the safety of particular probiotic strains.

One of the most recent systematic reviews identified 11,977 publications, of which 622 studies (included 24,615 participants using a probiotics) were included in the review. Based on reported adverse events, randomized controlled trials showed no statistically significantly increased relative risk of the over all number of experienced adverse events (Relative risk (RR) = 1.00; 95% Confidence interval (CI): 0.93, 1.07, p = 0.999); gastrointestinal; infections; or other adverse events, including serious adverse events (RR = 1.06; 95% CI: 0.97, 1.16; p = 0.201), associated with short-term probiotic use compared to control group participants; long-term effects are largely unknown. Case studies suggested that participants with compromised health are most likely to experience adverse events associated with probiotics. However, randomized control trials (RCTs) in medium-risk and critically ill participants did not report a statistically significantly increased risk of adverse events compared to control group participants. In conclusion authors of this analysis state, that the available evidence in RCTs does not indicate an increased risk; however, rare adverse events are difficult to assess. However, despite the substantial number of publications, the current literature is not well equipped to answer questions on the safety of probiotic interventions with confidence, especially in group of critically ill patients. Nevertheless, in specific probiotics group, as lactobacilli and bifidobacteria, some authors report that current evidence suggests, that the risk of infection with these probiotic groups is similar to that of infection with commensal strains and though consumption of such products presents a negligible risk to consumers, including immunocompromised hosts. Moreover, this potential risk needs to be always considered alongside any potential benefit. Despite limited data, it seems that probiotic bacteria as live microorganisms could be safely administered even in setting of neutropenia. Future research should focus on selection of most effective and safe probiotic strains and their combinations, and/or administration of probiotics with prebiotics to increase their success in maintaining colonization resistance and in prevention of the adverse events of anticancer treatment.

In a comparable study phase I. probiotic strain was applied to 11 cancer patients to evaluate their benefits and safety. Subsequently, 14 patients with acute myeloid leukemia treated with chemotherapy were enrolled in phase II. None of reported febrile episodes was induced by probiotic strain and no severe adverse events were recorded. Despite limited number of patients, this was the first direct evidence of the safety of probiotics in patients receiving chemotherapy.

One of the causes of failed efficacy of probiotics in the prevention of febrile neutropenia may be the presence of other entries of infection such as central venous catheters. Also, the efficiency of colonization, mucosal damage due to chemotherapy dose and specific probiotic strain may be the causes of this. Another reason may be the inability of one probiotic strain to compensate all changes in the intestinal microflora induced by chemotherapy. One way to solve this problem may be use of combination of multiple probiotic strains. Appropriate selection of strains is required, cause they must not behave antagonistically to each other. Other option is to use combination of prebiotics with probiotics. This can lead not only to acceleration of gut colonization by probiotics, but also to stimulation of endogenous flora growth, which may enhance colonization resistance at another level.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed cancer disease prior to initiation of chemotherapy
* Eastern Cooperative Oncology Group performance status = 0-1
* informed consent has to be given by patients, respectively their legal representatives
* age between 6 months to 19 years
* must be afebrile and no other signs of infection at least 24 hours before starting of prophylaxis
* must not taking other probiotic or prebiotic preparations or discontinued their use more than 14 days ago

Exclusion Criteria:

* impossibility of oral intake
* receiving any other type of experimental prophylaxis
* estimated survival time of less than 4 weeks
* allogeneic or autologous bone marrow transplantation
* inflammatory bowel disease

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-07; Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in the incidence of febrile neutropenia episodes | 3 months
  Febrile neutropenia is defined as an oral temperature >38.3°C or two consecutive readings of >38.0°C sustained for more than 1 hour and an absolute neutrophil count <0.5 × 109/l, or expected to fall below 0.5 × 109/l in the next 48-hour period

SECONDARY OUTCOMES:
Safety evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 3 months
  Safety will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03_2010-06-14_QuickReference_8.5x11.pdf
Reduction of the total duration of febrile neutropenia | 3 months
  Febrile neutropenia is defined as an oral temperature >38.3°C or two consecutive readings of >38.0°C sustained for more than 1 hour and an absolute neutrophil count <0.5 × 109/l, or expected to fall below 0.5 × 109/l in the next 48-hour period
Time period to first febrile episode | 3 months
Reduction in the number of septic complications requiring intensive care | 3 months
Reduction in the number of infectious episodes outside the period of neutropenia | 3 months
Reduction in the incidence of diarrhea and enterocolitis episodes related to chemotherapy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Holec, MD, PhD, Principal Investigator — University Children's Hospital Banska Bystrica; Michal Mego, MD, PhD, Principal Investigator — Comenius University and National Cancer Institute; Pavel Bician, MD, Study Chair — University Children's Hospital Banska Bystrica; Vladimir Zajac, RNDr, Study Chair — Slovak Academy of Sciences
Locations (1):
- University Children's Hospital Banska Bystrica, Banská Bystrica, Slovakia

REFERENCES:
- [Background] Cole GT, Halawa AA, Anaissie EJ. The role of the gastrointestinal tract in hematogenous candidiasis: from the laboratory to the bedside. Clin Infect Dis. 1996 May;22 Suppl 2:S73-88. doi: 10.1093/clinids/22.supplement_2.s73. PMID 8722833
- [Background] Klastersky J. A review of chemoprophylaxis and therapy of bacterial infections in neutropenic patients. Diagn Microbiol Infect Dis. 1989 Jul-Aug;12(4 Suppl):201S-207S. doi: 10.1016/0732-8893(89)90137-5. PMID 2686921
- [Background] Marshall JC. Gastrointestinal flora and its alterations in critical illness. Curr Opin Clin Nutr Metab Care. 1999 Sep;2(5):405-11. doi: 10.1097/00075197-199909000-00009. PMID 10589383
- [Background] Schimpff SC, Young VM, Greene WH, Vermeulen GD, Moody MR, Wiernik PH. Origin of infection in acute nonlymphocytic leukemia. Significance of hospital acquisition of potential pathogens. Ann Intern Med. 1972 Nov;77(5):707-14. doi: 10.7326/0003-4819-77-5-707. No abstract available. PMID 4628214
- [Background] Salva S, Marranzino G, Villena J, Aguero G, Alvarez S. Probiotic Lactobacillus strains protect against myelosuppression and immunosuppression in cyclophosphamide-treated mice. Int Immunopharmacol. 2014 Sep;22(1):209-21. doi: 10.1016/j.intimp.2014.06.017. Epub 2014 Jun 24. PMID 24975836
- [Background] Satonaka K, Ohashi K, Nohmi T, Yamamoto T, Abe S, Uchida K, Yamaguchi H. Prophylactic effect of Enterococcus faecalis FK-23 preparation on experimental candidiasis in mice. Microbiol Immunol. 1996;40(3):217-22. doi: 10.1111/j.1348-0421.1996.tb03337.x. PMID 8934676
- [Background] Shida K, Nomoto K. Probiotics as efficient immunopotentiators: translational role in cancer prevention. Indian J Med Res. 2013 Nov;138(5):808-14. PMID 24434333
- [Background] Shida K, Nanno M, Nagata S. Flexible cytokine production by macrophages and T cells in response to probiotic bacteria: a possible mechanism by which probiotics exert multifunctional immune regulatory activities. Gut Microbes. 2011 Mar-Apr;2(2):109-14. doi: 10.4161/gmic.2.2.15661. Epub 2011 Mar 1. PMID 21637028
- [Background] Perdigon G, Alvarez S, Rachid M, Aguero G, Gobbato N. Immune system stimulation by probiotics. J Dairy Sci. 1995 Jul;78(7):1597-606. doi: 10.3168/jds.S0022-0302(95)76784-4. PMID 7593855
- [Background] Marin ML, Tejada-Simon MV, Lee JH, Murtha J, Ustunol Z, Pestka JJ. Stimulation of cytokine production in clonal macrophage and T-cell models by Streptococcus thermophilus: comparison with Bifidobacterium sp. and Lactobacillus bulgaricus. J Food Prot. 1998 Jul;61(7):859-64. doi: 10.4315/0362-028x-61.7.859. PMID 9678170
- [Background] Neumann E, Oliveira MA, Cabral CM, Moura LN, Nicoli JR, Vieira EC, Cara DC, Podoprigora GI, Vieira LQ. Monoassociation with Lactobacillus acidophilus UFV-H2b20 stimulates the immune defense mechanisms of germfree mice. Braz J Med Biol Res. 1998 Dec;31(12):1565-73. doi: 10.1590/s0100-879x1998001200009. PMID 9951553
- [Background] Fuller R. Probiotics in man and animals. J Appl Bacteriol. 1989 May;66(5):365-78. PMID 2666378
- [Background] Gibson GR, Roberfroid MB. Dietary modulation of the human colonic microbiota: introducing the concept of prebiotics. J Nutr. 1995 Jun;125(6):1401-12. doi: 10.1093/jn/125.6.1401. PMID 7782892
- [Background] Resta-Lenert S, Barrett KE. Live probiotics protect intestinal epithelial cells from the effects of infection with enteroinvasive Escherichia coli (EIEC). Gut. 2003 Jul;52(7):988-97. doi: 10.1136/gut.52.7.988. PMID 12801956
- [Background] Vandenplas Y. Bacteria and yeasts in the treatment of acute and chronic infectious diarrhea. Part I. Bacteria. Clin Microbiol Infect. 1999 Jun;5(6):299-307. doi: 10.1111/j.1469-0691.1999.tb00148.x. PMID 11856274
- [Background] Apas AL, Gonzalez SN, Arena ME. Potential of goat probiotic to bind mutagens. Anaerobe. 2014 Aug;28:8-12. doi: 10.1016/j.anaerobe.2014.04.004. Epub 2014 Apr 29. PMID 24785349
- [Background] Mego M, Holec V, Drgona L, Hainova K, Ciernikova S, Zajac V. Probiotic bacteria in cancer patients undergoing chemotherapy and radiation therapy. Complement Ther Med. 2013 Dec;21(6):712-23. doi: 10.1016/j.ctim.2013.08.018. Epub 2013 Sep 1. PMID 24280481
- [Background] Redman MG, Ward EJ, Phillips RS. The efficacy and safety of probiotics in people with cancer: a systematic review. Ann Oncol. 2014 Oct;25(10):1919-1929. doi: 10.1093/annonc/mdu106. Epub 2014 Mar 11. PMID 24618152
- [Background] Sazawal S, Hiremath G, Dhingra U, Malik P, Deb S, Black RE. Efficacy of probiotics in prevention of acute diarrhoea: a meta-analysis of masked, randomised, placebo-controlled trials. Lancet Infect Dis. 2006 Jun;6(6):374-82. doi: 10.1016/S1473-3099(06)70495-9. PMID 16728323
- [Background] Isolauri E, Juntunen M, Rautanen T, Sillanaukee P, Koivula T. A human Lactobacillus strain (Lactobacillus casei sp strain GG) promotes recovery from acute diarrhea in children. Pediatrics. 1991 Jul;88(1):90-7. PMID 1905394
- [Background] Born P, Lersch C, Zimmerhackl B, Classen M. [The Saccharomyces boulardii therapy of HIV-associated diarrhea]. Dtsch Med Wochenschr. 1993 May 21;118(20):765. No abstract available. German. PMID 8500427
- [Background] Saint-Marc T, Rossello-Prats L, Touraine JL. [Efficacy of Saccharomyces boulardii in the treatment of diarrhea in AIDS]. Ann Med Interne (Paris). 1991;142(1):64-5. No abstract available. French. PMID 2048880
- [Background] Hasegawa T, Kanasugi H, Hidaka M, Yamamoto T, Abe S, Yamaguchi H. Effect of orally administered heat-killed Enterococcus Faecalis FK-23 preparation on neutropenia in dogs treated with cyclophosphamide. Int J Immunopharmacol. 1996 Feb;18(2):103-12. doi: 10.1016/0192-0561(96)00001-x. PMID 8799360
- [Background] Vanderhoof JA, Young R. Probiotics in the United States. Clin Infect Dis. 2008 Feb 1;46 Suppl 2:S67-72; discussion S144-51. doi: 10.1086/523339. PMID 18181726
- [Background] Swenson JM, Facklam RR, Thornsberry C. Antimicrobial susceptibility of vancomycin-resistant Leuconostoc, Pediococcus, and Lactobacillus species. Antimicrob Agents Chemother. 1990 Apr;34(4):543-9. doi: 10.1128/AAC.34.4.543. PMID 2344161
- [Background] Handwerger S, Pucci MJ, Volk KJ, Liu J, Lee MS. Vancomycin-resistant Leuconostoc mesenteroides and Lactobacillus casei synthesize cytoplasmic peptidoglycan precursors that terminate in lactate. J Bacteriol. 1994 Jan;176(1):260-4. doi: 10.1128/jb.176.1.260-264.1994. PMID 8282706
- [Background] Klein G, Pack A, Bonaparte C, Reuter G. Taxonomy and physiology of probiotic lactic acid bacteria. Int J Food Microbiol. 1998 May 26;41(2):103-25. doi: 10.1016/s0168-1605(98)00049-x. PMID 9704860
- [Background] Charteris WP, Kelly PM, Morelli L, Collins JK. Antibiotic susceptibility of potentially probiotic Lactobacillus species. J Food Prot. 1998 Dec;61(12):1636-43. doi: 10.4315/0362-028x-61.12.1636. PMID 9874341
- [Background] Salminen S, von Wright A, Morelli L, Marteau P, Brassart D, de Vos WM, Fonden R, Saxelin M, Collins K, Mogensen G, Birkeland SE, Mattila-Sandholm T. Demonstration of safety of probiotics -- a review. Int J Food Microbiol. 1998 Oct 20;44(1-2):93-106. doi: 10.1016/s0168-1605(98)00128-7. PMID 9849787
- [Background] Tynkkynen S, Singh KV, Varmanen P. Vancomycin resistance factor of Lactobacillus rhamnosus GG in relation to enterococcal vancomycin resistance (van) genes. Int J Food Microbiol. 1998 Jun 16;41(3):195-204. doi: 10.1016/s0168-1605(98)00051-8. PMID 9706787
- [Background] Ahn C, Collins-Thompson D, Duncan C, Stiles ME. Mobilization and location of the genetic determinant of chloramphenicol resistance from Lactobacillus plantarum caTC2R. Plasmid. 1992 May;27(3):169-76. doi: 10.1016/0147-619x(92)90018-6. PMID 1513874
- [Background] Gevers D, Danielsen M, Huys G, Swings J. Molecular characterization of tet(M) genes in Lactobacillus isolates from different types of fermented dry sausage. Appl Environ Microbiol. 2003 Feb;69(2):1270-5. doi: 10.1128/AEM.69.2.1270-1275.2003. PMID 12571056
- [Background] Ishiwa H, Iwata S. Drug resistance plasmids in Lactobacillus fermetum. J Gen Appl Microbiol 1980; 26:71-4.
- [Background] Fons M, Hege T, Ladire M, Raibaud P, Ducluzeau R, Maguin E. Isolation and characterization of a plasmid from Lactobacillus fermentum conferring erythromycin resistance. Plasmid. 1997;37(3):199-203. doi: 10.1006/plas.1997.1290. PMID 9200223
- [Background] Tannock GW, Luchansky JB, Miller L, Connell H, Thode-Andersen S, Mercer AA, Klaenhammer TR. Molecular characterization of a plasmid-borne (pGT633) erythromycin resistance determinant (ermGT) from Lactobacillus reuteri 100-63. Plasmid. 1994 Jan;31(1):60-71. doi: 10.1006/plas.1994.1007. PMID 8171126
- [Background] Morelli L, Wright AV. Probiotic bacteria and transferable antibiotic resistance-safety aspects. Demonstration of the Nutritional Functionality of Probiotic Foods News Letter 1997; 2:9-14.
- [Background] Saarela M, Mogensen G, Fonden R, Matto J, Mattila-Sandholm T. Probiotic bacteria: safety, functional and technological properties. J Biotechnol. 2000 Dec 28;84(3):197-215. doi: 10.1016/s0168-1656(00)00375-8. PMID 11164262
- [Background] Salyers AA, Gupta A, Wang Y. Human intestinal bacteria as reservoirs for antibiotic resistance genes. Trends Microbiol. 2004 Sep;12(9):412-6. doi: 10.1016/j.tim.2004.07.004. PMID 15337162
- [Background] Mathur S, Singh R. Antibiotic resistance in food lactic acid bacteria--a review. Int J Food Microbiol. 2005 Dec 15;105(3):281-95. doi: 10.1016/j.ijfoodmicro.2005.03.008. Epub 2005 Nov 8. PMID 16289406
- [Background] Gasser S. Safety of lactic acid bacteria and their occurrence in human clinical infection. Bull Inst Pasteur 1994; 92:45-67.
- [Background] Fruchart C, Salah A, Gray C, Martin E, Stamatoullas A, Bonmarchand G, Lemeland JF, Tilly H. Lactobacillus species as emerging pathogens in neutropenic patients. Eur J Clin Microbiol Infect Dis. 1997 Sep;16(9):681-4. doi: 10.1007/BF01708560. PMID 9352263
- [Background] Land MH, Rouster-Stevens K, Woods CR, Cannon ML, Cnota J, Shetty AK. Lactobacillus sepsis associated with probiotic therapy. Pediatrics. 2005 Jan;115(1):178-81. doi: 10.1542/peds.2004-2137. PMID 15629999
- [Background] Kalima P, Masterton RG, Roddie PH, Thomas AE. Lactobacillus rhamnosus infection in a child following bone marrow transplant. J Infect. 1996 Mar;32(2):165-7. doi: 10.1016/s0163-4453(96)91622-9. PMID 8708379
- [Background] Schlegel L, Lemerle S, Geslin P. Lactobacillus species as opportunistic pathogens in immunocompromised patients. Eur J Clin Microbiol Infect Dis. 1998 Dec;17(12):887-8. doi: 10.1007/s100960050216. No abstract available. PMID 10052559
- [Background] Saxelin M, Chuang NH, Chassy B, Rautelin H, Makela PH, Salminen S, Gorbach SL. Lactobacilli and bacteremia in southern Finland, 1989-1992. Clin Infect Dis. 1996 Mar;22(3):564-6. doi: 10.1093/clinids/22.3.564. PMID 8852980
- [Background] Ouwehand AC, Saxelin M, Salminen S. Phenotypic differences between commercial Lactobacillus rhamnosus GG and L. rhamnosus strains recovered from blood. Clin Infect Dis. 2004 Dec 15;39(12):1858-60. doi: 10.1086/425741. Epub 2004 Nov 19. PMID 15578412
- [Background] Kirjavainen PV, Tuomola EM, Crittenden RG, Ouwehand AC, Harty DW, Morris LF, Rautelin H, Playne MJ, Donohue DC, Salminen SJ. In vitro adhesion and platelet aggregation properties of bacteremia-associated lactobacilli. Infect Immun. 1999 May;67(5):2653-5. doi: 10.1128/IAI.67.5.2653-2655.1999. PMID 10225937
- [Background] Berg RD. Bacterial translocation from the gastrointestinal tract. Trends Microbiol. 1995 Apr;3(4):149-54. doi: 10.1016/s0966-842x(00)88906-4. PMID 7613757
- [Background] Berg RD. Translocation and the indigenous gut flora. In: FullerR, editor. Probiotics: the scientific basis. London: Chapman &Hall 1992; 55-85.83.
- [Background] Pavan S, Desreumaux P, Mercenier A. Use of mouse models to evaluate the persistence, safety, and immune modulation capacities of lactic acid bacteria. Clin Diagn Lab Immunol. 2003 Jul;10(4):696-701. doi: 10.1128/cdli.10.4.696-701.2003. PMID 12853407
- [Background] Chiva M, Soriano G, Rochat I, Peralta C, Rochat F, Llovet T, Mirelis B, Schiffrin EJ, Guarner C, Balanzo J. Effect of Lactobacillus johnsonii La1 and antioxidants on intestinal flora and bacterial translocation in rats with experimental cirrhosis. J Hepatol. 2002 Oct;37(4):456-62. doi: 10.1016/s0168-8278(02)00142-3. PMID 12217598
- [Background] Shu Q, Gill HS. Immune protection mediated by the probiotic Lactobacillus rhamnosus HN001 (DR20) against Escherichia coli O157:H7 infection in mice. FEMS Immunol Med Microbiol. 2002 Sep 6;34(1):59-64. doi: 10.1111/j.1574-695X.2002.tb00603.x. PMID 12208607
- [Background] Romond MB, Haddou Z, Mielcareck C, Romond C. Bifidobacteria and human health: regulatory effect of indigenous bifidobacteria on Escherichia coli intestinal colonization. Anaerobe. 1997 Apr-Jun;3(2-3):131-6. doi: 10.1006/anae.1997.0089. PMID 16887577
- [Background] Durand JM, Rousseau MC, Gandois JM, Kaplanski G, Mallet MN, Soubeyrand J. Streptococcus lactis septicemia in a patient with chronic lymphocytic leukemia. Am J Hematol. 1995 Sep;50(1):64-5. doi: 10.1002/ajh.2830500116. No abstract available. PMID 7668230
- [Background] Cairoli R, Marenco P, Perego R, de Cataldo F. Saccharomyces cerevisiae fungemia with granulomas in the bone marrow in a patient undergoing BMT. Bone Marrow Transplant. 1995 May;15(5):785-6. PMID 7670407
- [Background] Salminen MK, Tynkkynen S, Rautelin H, Saxelin M, Vaara M, Ruutu P, Sarna S, Valtonen V, Jarvinen A. Lactobacillus bacteremia during a rapid increase in probiotic use of Lactobacillus rhamnosus GG in Finland. Clin Infect Dis. 2002 Nov 15;35(10):1155-60. doi: 10.1086/342912. Epub 2002 Oct 21. PMID 12410474
- [Background] Wolf BW, Wheeler KB, Ataya DG, Garleb KA. Safety and tolerance of Lactobacillus reuteri supplementation to a population infected with the human immunodeficiency virus. Food Chem Toxicol. 1998 Dec;36(12):1085-94. doi: 10.1016/s0278-6915(98)00090-8. PMID 9862651
- [Background] Cunningham-Rundles S, Ahrne S, Bengmark S, Johann-Liang R, Marshall F, Metakis L, Califano C, Dunn AM, Grassey C, Hinds G, Cervia J. Probiotics and immune response. Am J Gastroenterol. 2000 Jan;95(1 Suppl):S22-5. doi: 10.1016/s0002-9270(99)00813-8. PMID 10634225
- [Background] Hempel S, Newberry S, Ruelaz A, Wang Z, Miles JN, Suttorp MJ, Johnsen B, Shanman R, Slusser W, Fu N, Smith A, Roth B, Polak J, Motala A, Perry T, Shekelle PG. Safety of probiotics used to reduce risk and prevent or treat disease. Evid Rep Technol Assess (Full Rep). 2011 Apr;(200):1-645. PMID 23126627
- [Background] Agostoni C, Axelsson I, Braegger C, Goulet O, Koletzko B, Michaelsen KF, Rigo J, Shamir R, Szajewska H, Turck D, Weaver LT; ESPGHAN Committee on Nutrition. Probiotic bacteria in dietetic products for infants: a commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2004 Apr;38(4):365-74. doi: 10.1097/00005176-200404000-00001. No abstract available. PMID 15085012
- [Background] Naidu AS, Bidlack WR, Clemens RA. Probiotic spectra of lactic acid bacteria (LAB). Crit Rev Food Sci Nutr. 1999 Jan;39(1):13-126. doi: 10.1080/10408699991279187. PMID 10028126
- [Background] Borriello SP, Hammes WP, Holzapfel W, Marteau P, Schrezenmeir J, Vaara M, Valtonen V. Safety of probiotics that contain lactobacilli or bifidobacteria. Clin Infect Dis. 2003 Mar 15;36(6):775-80. doi: 10.1086/368080. Epub 2003 Mar 5. PMID 12627362
- [Background] Hammerman C, Bin-Nun A, Kaplan M. Safety of probiotics: comparison of two popular strains. BMJ. 2006 Nov 11;333(7576):1006-8. doi: 10.1136/bmj.39010.630799.BE. No abstract available. PMID 17095783
- [Background] Mego M, Ebringer L, Drgona L, Mardiak J, Trupl J, Greksak R, Nemova I, Oravcova E, Zajac V, Koza I. Prevention of febrile neutropenia in cancer patients by probiotic strain Enterococcus faecium M-74. Pilot study phase I. Neoplasma. 2005;52(2):159-64. PMID 15800715
- [Background] Mego M, Koncekova R, Mikuskova E, Drgona L, Ebringer L, Demitrovicova L, Nemova I, Trupl J, Mardiak J, Koza I, Zajac V. Prevention of febrile neutropenia in cancer patients by probiotic strain Enterococcus faecium M-74. Phase II study. Support Care Cancer. 2006 Mar;14(3):285-90. doi: 10.1007/s00520-005-0891-7. Epub 2005 Sep 21. PMID 16175356